CLINICAL TRIAL: NCT06174727
Title: Outcomes of Intra-arterial and Endosaccular Flow Diverters for Treatment of Intracranial Aneurysms - International Registry of Intra-arterial and Endosaccular Flow Diverters (IRF)
Brief Title: International Registry of Intra-arterial and Endosaccular Flow Diverters (IRF)
Acronym: IRF
Status: Recruiting | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Mayo Clinic (Other); Simpson Memorial Research Institute (Other); Geisinger Health (Unknown); University at Buffalo (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-15177
Record Dates: First submitted 2023-12-05; First posted 2023-12-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Aneurysm
Keywords: Endovascular; Registry; Flow Diverter Stents; Endosaccular Flow Disruptors; Flow Diversion
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter retrospective cohort study aims to evaluate and compare the technical performance, safety, and clinical outcomes of intracranial aneurysms treated with flow diverter stents and endosaccular flow disruptors.

DETAILED DESCRIPTION:
Flow diverters and endosaccular flow disruptors used for the treatment of intracranial aneurysms exhibit distinct procedural and clinical outcomes, with potential differences in device-specific parameters such as procedure time, radiation exposure, adjunct device requirements, and long-term angiographic success. Since the completion of the Pipeline Embolization Device (PED) for the Intracranial Treatment of Aneurysms trial, the field of flow diversion has undergone continuous evolution with the development and approval of several devices. While these devices share a similar mechanism for aneurysm occlusion, their design and delivery systems can vary significantly. Various studies have demonstrated a promising safety and efficacy profile; however, the available data for a direct comparison of the technical and clinical outcomes between these devices remains limited.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or older)
* Underwent endovascular treatment with one of the following devices:

  a. Endoluminal Flow Diverter Stents: i. Pipeline Flex (Covidien, California, USA) ii. Pipeline Flex with Shield Technology (Covidien) iii. Surpass Streamline (Stryker Neurovascular, California, USA) iv. Surpass Evolve (Stryker) v. Silk flow diverter (Balt Extrusion, Montmorency, France) vi. Flow-Redirection Intraluminal Device (FRED; MicroVention) vii. Flow-Redirection Intraluminal Device X (FRED X; MicroVention) viii. p64 Flow Modulation Device (phenox GmbH) ix. Endovascular clip system (eCLIPs) (eCLIPsTM, eVasc Neurovascular, Vancouver, BC, Canada)

  b. Intrasaccular Flow Disruptors: i. Woven EndoBridge (WEB; MicroVention) ii. Luna/Artisse System (Medtronic) iii. Medina Embolic Device (Medtronic) iv. Contour Neurovascular System (Cerus Endovascular) v. Neqstent Coil Assisted Flow Diverter (Cerus Endovascular) vi. pCONus and pCANvas (phenox GmbH) vii. Nexus Aneurysm Embolization System (EndoStream Medical) viii. CITADEL™ Embolization Device (Balt, USA)
* Complete medical records and follow-up data available

Exclusion Criteria:

* Incomplete procedural or follow-up records
* Non-flow-diverter or non-flow-disruptor treatments (e.g., coiling-only cases)
* Aneurysms treated with investigational devices not listed within Inclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial aneurysms who underwent endovascular treatment with flow diverter stents or endosaccular flow disruptors
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Technical Success | Periprocedurally, up to 24 hours
  Technical Success will be determined by successful deployment of the flow diverter stent or endosaccular flow disruptors. A dichotomous determination (i.e., Yes/No) will be made and summarized for this study.
Procedural Complications following placement | From the time of the procedure up to 1 month post treatment
  Procedural complications will be identified as the number of instances of the following adverse clinical events: In-stent Thrombosis/Stenosis; Ischemic complications (Transient Ischemic Attack/Stroke), Intracerebral hemorrhage, Aneurysm rupture, and Vessel occlusion due to flow diverter stent or endosaccular flow disruptor placement.
Clinical Outcomes at Discharge | Upon study discharge, up to 4 weeks
  Clinical outcomes at discharge will be assessed using the modified Rankin Scale (mRS) for neurologic disability. The mRS is a 6-point disability scale with possible scores ranging from 0-5. mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Higher scores are generally associated with less favorable outcomes. For this study patients with an mRS score of 0-2 will be determined to have had a "favorable" outcome to the procedure and patients with an mRS score of 3-5 will have been determined to have had an "unfavorable" outcome.
Clinical Outcomes at last available Follow-up | Up to 24 months post procedure
  Clinical outcomes at last available follow-up will be assessed using a variant of the modified Rankin Scale (mRS) for neurologic disability. The classic mRS is a 6-point disability scale with possible scores ranging from 0-5. mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Higher scores are generally associated with less favorable outcomes. For this study patients with an mRS score of 0-2 will be determined to have had a "favorable" outcome to the procedure and patients with an mRS score of 3-5 will have been determined to have had an "unfavorable" outcome. Scoring will also include a 6 to identify patients who have expired.
Immediate Angiographic Outcomes at Discharge - O'Kelly-Marotta (OKM) grading scale | Upon study discharge, up to 4 weeks
  Immediate Angiographic Outcomes at Discharge will be evaluated using the OKM grading scale. The OKM scale will be used to assess the degree of angiographic filling and in the setting of intracranial aneurysms which were treated by endovascular flow diversion. It is used to predict aneurysm closure over time. Patient outcomes will be stratified based on the following scale scores: Grade A: Total filling (>95% of aneurysm remained); Grade B: Subtotal filling (5-95% of aneurysm remained); Grade C: Entry remnant (<5% aneurysm remained); and Grade D: No filling (0% aneurysm remained). As such, the less aneurysm remnant the more favorable the angiographic outcome. The number/percentage of cases of each OKM Grade will be summarized.
Immediate Angiographic Outcomes at Discharge - Modified Raymond-Roy Classification (mRRC) | Upon study discharge, up to 4 weeks
  Immediate Angiographic Outcomes at Discharge will also be evaluated using mRRC categorization. mRRC categorization will be used to assess the degree of occlusion achieved when treating an intracranial aneurysm. It categorizes the level of residual contrast filling within an aneurysm after coiling. For purposes of this analysis, Class I will signify complete occlusion; Class II will signify Residual neck occlusion; Class IIIa will signify Residual aneurysm with contrast stasis; and Class IIIb will signify Residual aneurysm without contrast stasis. As such, it is an indicator of how effectively the aneurysm has been sealed off during treatment. The number/percentage of cases of each mRRC category will be summarized.
Immediate Angiographic Outcomes at Discharge - WEB Occlusion Scale (WOS) | Upon study discharge, up to 4 weeks
  Immediate Angiographic Outcomes at Discharge will be evaluated using the WOS grading scale. The WOS is a standardized angiographic assessment scale for reporting aneurysm occlusion achieved with endosaccular flow disruptors and can be employed to assess the adequacy of treatment. For purposes of this analysis, WOS Grade A will signify complete occlusion; WOS Grade B will signify Residual neck occlusion; and WOS Grade C will signify Residual aneurysm filling. The number/percentage of cases of each WOS grade category will be summarized.
Angiographic Outcomes at last available Follow-up - O'Kelly-Marotta (OKM) grading scale | Up to 24 months post procedure
  Immediate Angiographic Outcomes at Discharge will be evaluated using the OKM grading scale. The OKM scale will be used to assess the degree of angiographic filling and in the setting of intracranial aneurysms which were treated by endovascular flow diversion. It is used to predict aneurysm closure over time. Patient outcomes will be stratified based on the following scale scores: Grade A: Total filling (>95% of aneurysm remained); Grade B: Subtotal filling (5-95% of aneurysm remained); Grade C: Entry remnant (<5% aneurysm remained); and Grade D: No filling (0% aneurysm remained). As such, the less aneurysm remnant the more favorable the angiographic outcome. The number/percentage of cases of each OKM Grade will be summarized.
Angiographic Outcomes at last available Follow-up - Modified Raymond-Roy Classification (mRRC) | Up to 24 months post procedure
  Immediate Angiographic Outcomes at Discharge will also be evaluated using mRRC categorization. mRRC categorization will be used to assess the degree of occlusion achieved when treating an intracranial aneurysm. It categorizes the level of residual contrast filling within an aneurysm after coiling. For purposes of this analysis, Class I will signify complete occlusion; Class II will signify Residual neck occlusion; Class IIIa will signify Residual aneurysm with contrast stasis; and Class IIIb will signify Residual aneurysm without contrast stasis. As such, it is an indicator of how effectively the aneurysm has been sealed off during treatment. The number/percentage of cases of each mRRC category will be summarized.
Angiographic Outcomes at last available Follow-up - WEB Occlusion Scale (WOS) | Up to 24 months post procedure
  Immediate Angiographic Outcomes at Discharge will be evaluated using the WOS grading scale. The WOS is a standardized angiographic assessment scale for reporting aneurysm occlusion achieved with endosaccular flow disruptors and can be employed to assess the adequacy of treatment. For purposes of this analysis, WOS Grade A will signify complete occlusion; WOS Grade B will signify Residual neck occlusion; and WOS Grade C will signify Residual aneurysm filling. The number/percentage of cases of each WOS grade category will be summarized.

SECONDARY OUTCOMES:
Radiation Exposure | Periprocedurally, up to 4 hours
  Radiation exposure over the course of the procedure will be extracted and summarized. Radiation exposure will be evaluated based on relevant imaging system metrics used to calculate the total radiation dose delivered to the patient based on the fluoroscopy time and the area of the X-ray field exposed during the procedure. Flow diverter stents and endosaccular flow disruptors typically result in significantly lower radiation exposure compared to other endovascular techniques for treating brain aneurysms due to a reduction in fluoroscopy time and overall reduced radiation dose due to the streamlined nature of the procedures.
Procedure Duration | Periprocedurally, up to 4 hours
  The duration of procedure placement will be extracted and summarized. The duration of the procedure is influenced by the complexity of the aneurysm, the patient's anatomy, and the experience of the interventional radiologist and care team. Shorter procedure duration times are associated with more favorable outcomes.
Use of Adjunct Devices | Periprocedurally, up to 4 hours
  The use of adjunctive devices such as coils, stents or balloons to further enhance aneurysm occlusion of the flow diverter stent or to facilitate positioning and deployment of the endosaccular flow disruptor within the aneurysm sac during the procedure will be extracted and summarized. The number of adjunct devices will be extracted and summarized.
Recurrence of Aneurysm | 6 to 24 months post procedure
  The percentage of patients who experienced aneurysm recurrence will be extracted and summarized based on a binary (Yes/No) determination following retrospective record review. The span of time from initial treatment to recurrence will be assessed and summarized.
Aneurysm Retreatment | 6 to 24 months post procedure
  The percentage of patients who required retreatment for a recurrence of aneurysm will be extracted and summarized based on a binary (Yes/No) determination following retrospective record review. The span of time from initial treatment to retreatment will be assessed and summarized.

CONTACTS AND LOCATIONS:
Overall Officials: David Altschul, MD, Principal Investigator — Montefiore Medical Center
Locations (11):
- United States (10):
  - University of Miami, Coral Gables, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Sarasota Memorial Research Institute, Sarasota, Florida
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Munson Medical Center, Traverse City, Michigan
  - Robert Wood Johnson University, New Brunswick, New Jersey
  - University at Buffalo, Buffalo, New York
  - Montefiore Medical Center Department of Neurosurgery, The Bronx, New York
  - Geisinger Health, Danville, Pennsylvania
  - HCA Houston Healthcare Kingwood, Kingwood, Texas
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson PK, Lylyk P, Szikora I, Wetzel SG, Wanke I, Fiorella D. The pipeline embolization device for the intracranial treatment of aneurysms trial. AJNR Am J Neuroradiol. 2011 Jan;32(1):34-40. doi: 10.3174/ajnr.A2421. Epub 2010 Dec 9. PMID 21148256
- [Background] Hecker C, Broussalis E, Griessenauer CJ, Killer-Oberpfalzer M. A mini-review of intrasaccular flow diverters. J Neurointerv Surg. 2023 Jan;15(1):70-74. doi: 10.1136/neurintsurg-2021-018426. Epub 2022 May 17. PMID 35580985
- [Background] Colby GP, Lin LM, Caplan JM, Jiang B, Michniewicz B, Huang J, Tamargo RJ, Coon AL. Flow diversion of large internal carotid artery aneurysms with the surpass device: impressions and technical nuance from the initial North American experience. J Neurointerv Surg. 2016 Mar;8(3):279-86. doi: 10.1136/neurintsurg-2015-011769. Epub 2015 May 18. PMID 25987590
- [Background] Vivanco-Suarez J, Feigen C, Javed K, Dardick JM, Holland R, Mendez-Ruiz A, Ortega-Gutierrez S, Haranhalli N, Altschul DJ. Dataset on flow diversion procedures performed with the Pipeline Embolization Device, Pipeline Flex, and Surpass Streamline for intracranial aneurysms. Data Brief. 2022 May 21;42:108299. doi: 10.1016/j.dib.2022.108299. eCollection 2022 Jun. PMID 35669008
- [Background] Wakhloo AK, Lylyk P, de Vries J, Taschner C, Lundquist J, Biondi A, Hartmann M, Szikora I, Pierot L, Sakai N, Imamura H, Sourour N, Rennie I, Skalej M, Beuing O, Bonafe A, Mery F, Turjman F, Brouwer P, Boccardi E, Valvassori L, Derakhshani S, Litzenberg MW, Gounis MJ; Surpass Study Group. Surpass flow diverter in the treatment of intracranial aneurysms: a prospective multicenter study. AJNR Am J Neuroradiol. 2015 Jan;36(1):98-107. doi: 10.3174/ajnr.A4078. Epub 2014 Aug 14. PMID 25125666
- [Background] O'kelly CJ, Krings T, Fiorella D, Marotta TR. A novel grading scale for the angiographic assessment of intracranial aneurysms treated using flow diverting stents. Interv Neuroradiol. 2010 Jun;16(2):133-7. doi: 10.1177/159101991001600204. Epub 2010 Jul 19. PMID 20642887